CLINICAL TRIAL: NCT03177265
Title: Text Messaging to Engage and Retain Veterans in Smoking Cessation Counseling
Acronym: TiMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: IIR 15-297
Record Dates: First submitted 2017-05-31; First posted 2017-06-06 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Nicotine Dependence
Keywords: nicotine dependence; tobacco cessation
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use Cessation

STUDY DESIGN:
Intervention Model Description: The investigators will first randomize each Veteran, stratified by site, to: a) Text-to-Engage vs. standard Proactive Outreach (PrO). For those who enroll in counseling, the investigators will then randomize them to: b) Text-to-Enhance + Telephone Counseling vs. Telephone Counseling alone (TelC). Primary outcomes will be the rate of enrollment in counseling and cotinine-verified quit rate at 12 months.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Text to Engage (Experimental): This group will get 8 text messages that target common misperceptions around quitting and use of quit services prior to receiving the first counseling phone call.
  Interventions: Behavioral: Text messaging prior to first counseling call
- Mail Notice (Other): This group will only get a mailing indicating that they will receive a call from a quitline counseling in two weeks.
  Interventions: Behavioral: Mail Notice
- Text to Enhance (Experimental): Text-to-Enhance condition will receive SMS appointment reminders for telephone counseling appointments and 5 texts per week with tips and suggestions for quitting for a duration of 8 weeks.
  Interventions: Behavioral: Text-to-Enhance
- Telephone Counseling (Active Comparator): Telephone counseling condition will receive standard 8 weeks of telephone counseling only.
  Interventions: Behavioral: Telephone Counseling

INTERVENTIONS:
Behavioral: Text messaging prior to first counseling call — This is the first randomization (text to engage vs. mailed notice). Patients randomized to this condition will receive up to 8 text messages prior to the first counseling phone call to provide education regarding cessation treatment.
  Other Names: Text to Engage.
  Arms: Text to Engage
Behavioral: Text-to-Enhance — Two weeks following receipt of the letter (PrO condition) or upon completion of the engagement text messages (Text-to-Engage condition) a counselor trained in motivational interviewing and smoking cessation treatment will phone participants. The Text-to-Enhance condition will receive SMS appointment reminders for telephone counseling appointments and 5 texts per week with tips and suggestions for quitting for a duration of 8 weeks. The telephone counseling condition will receive standard 8 weeks of telephone counseling only.
  Arms: Text to Enhance
Behavioral: Mail Notice — This is the first randomization (text to engage vs. mailed notice). Patients randomized to this condition will receive a notice in the mail that they will receive a phone call in about 2 weeks to offer telephone cessation treatment.
  Arms: Mail Notice
Behavioral: Telephone Counseling — Two weeks following receipt of the mailed notice or upon completion of the engagement text messages (Text-to-Engage condition) a counselor trained in motivational interviewing and smoking cessation treatment will phone participants. The Text-to-Enhance condition will receive SMS appointment reminders for telephone counseling appointments and 5 texts per week with tips and suggestions for quitting for a duration of 8 weeks. The telephone counseling condition will receive standard 8 weeks of telephone counseling only.
  Arms: Telephone Counseling

SUMMARY:
Tobacco-related diseases account for a significant portion of all VA healthcare costs and are a detriment to the health and quality of life of our Veterans. Despite progress in instituting tobacco screenings and treatment referral, most Veterans still do not receive the most effective strategy to help them quit smoking - pharmacotherapy combined with behavioral coaching. This study builds on findings from population health and mobile interventions to help more Veterans receive evidence-based tobacco treatment. The investigators propose to test the effect of two types of text messaging in combination with telephone cessation counseling: 1) pre-counseling text messages to increase enrollment in counseling, and 2) ongoing texts for those who start counseling that provide appointment reminders and support between sessions to increase adherence to counseling. This study supports multiple goals of the VA's Blueprint for Excellence. Results will directly inform decision-making and population-based care models for tobacco treatment.

DETAILED DESCRIPTION:
Tobacco use remains the number one cause of premature death and morbidity in the United States, and tobacco-related diseases account for 24% of all VA healthcare costs. The VA has been a leader in addressing tobacco use, having implemented annual tobacco screening and made pharmacotherapy readily available. However, one of the most cost-effective services - telephone quit lines - remain highly underused. Few Veterans enroll in telephone counseling to help them quit smoking, and among Veterans who begin telephone counseling, few complete a full course. The advent of electronic health records (EHRs) has enabled new strategies for ensuring that patients receive preventive services. These methods can reduce provider burden and close gaps in systems of care. The investigators' research team has conducted numerous studies using EHRs to identify smokers and proactively reach out to coordinate telephone tobacco treatment. While the investigators have successfully implemented this approach, the overall enrollment rates for counseling remain low and the majority of smokers complete only one counseling session. Therefore, the investigators propose to test novel mHealth strategies for promoting enrollment in and adherence to telephone counseling. The Specific Aims are to: 1) Conduct a sequentially randomized trail to estimate the effectiveness of text messaging for increasing enrollment in and adherence to telephone tobacco treatment, 2) Compare rates of tobacco cessation between patients who received and did not receive text messaging during treatment, and 3) Evaluate patient experiences with these interventions. Using the VA EHR, the investigators will identify N=3,600 smokers at two VA sites. All identified smokers will be mailed an introductory packet with information about the study. Patients who consent will be randomized to standard telephone outreach for counseling or to receive 8 educational texts to counter barriers of participating in counseling prior to telephone outreach. Patients who enroll in tobacco treatment will then be randomized to receive standard telephone counseling or to also receive appointment reminders and supportive texts throughout the 8-week counseling period. The investigators hypothesize that these approaches will increase the rate of enrollment in telephone tobacco cessation and 12-month biochemically validated abstinence (primary outcomes) over standard telephone counseling approaches. The investigators will also assess patient experiences with each texting protocol. The investigators' overarching goal is to investigative innovative mHealth strategies for increasing Veteran use of telephone-based tobacco cessation counseling and to improve quit rates. This research, exploring both population-based outreach and text messaging, advances multiple goals set forth by the VA's Blueprint for Excellence. Results will have direct implications to inform decision-making and population-based care models for tobacco treatment.

ELIGIBILITY:
Inclusion Criteria:

* Current smoker (i.e., positive tobacco use in past 6 months)
* Veteran 18 years or older
* Cell phone number listed the medical record

Exclusion Criteria:

* ICD 9 diagnosis of dementia (excluded during data abstraction process)
* Does not speak English
* No mailing address (necessary to mail out initial study materials)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
cotinine-verified quit rate | 12 months
  Tobacco cessation will be verified via oral swab cotinine.

SECONDARY OUTCOMES:
Rate of enrollment in telephone counseling | at completion of recruitment, average of 1 year
  This will be calculated from the number who enroll in counseling divided by 1,800 separately for each study condition.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Krebs, PhD, Principal Investigator — Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY
Locations (2):
- United States (2):
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York

IPD SHARING:
Plan to Share IPD: No
We will prepare multiple manuscripts to be submitted to peer-review journals summarizing our findings. We will disseminate our study findings through several additional channels:
  * Traditional Dissemination - We will send a study report to each facility's leadership, including the medical center Director and ACOS of Research, for their review. We will also publish findings in relevant journals
  * We will submit one or more abstracts to the annual HSR&D meeting as well as other gatherings of health service professionals.
  * VA Office of Connected Health - We will share our study findings with the Office of Connected Health in order to provide data regarding potential uses of efficacy of the technologies they are supporting.
  Access to data will be made available to any researcher wishing to analyze data with a research protocol approved by the IRB and with a data use agreement approved by the PO and ISO at our facility.